CLINICAL TRIAL: NCT05668624
Title: Sustainable Household Energy Adoption in Rwanda (SHEAR): Promoting Rural Health With Solar and Natural Gas
Brief Title: Sustainable Household Energy Adoption in Rwanda (SHEAR)
Acronym: SHEAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2219; R01ES029995 (NIH)
Record Dates: First submitted 2022-12-07; First posted 2022-12-30 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Blood Pressure; Lung Function

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Full Subsidy Arm (Experimental): This arm receives free LPG and stove for cooking following the baseline measures, for the duration of the 3-year follow-up period. For those households in Government of Rwanda designated areas for solar microgrids, this arm will also be connected to and provided free access to solar electricity for lighting.
  Interventions: Other: Clean household energy
- Control Arm (No Intervention): This arm will remain using traditional forms of energy for cooking and lighting.
- Discount Subsidy Arm (Experimental): This arm will be randomized to a discounted price (at baseline and every 6-months during the 3-year study) for solar electricity (in areas marker for solar grids by the Government of Rwanda) and LPG gas in a pay-as-you-go (PAYG) service model (i.e., pre-pay an affordable amount through mobile money, a common form of currency transactions in Rwanda). For example, this arm will be asked to cook as normal and decide whether or not to cook with the discounted LPG or their traditional stove (i.e., they will not be required to pay for LPG).
  Interventions: Other: Clean household energy

INTERVENTIONS:
Other: Clean household energy — LPG stoves/fuel for cooking and solar electricity for lighting
  Arms: Discount Subsidy Arm; Full Subsidy Arm

SUMMARY:
Investigators will conduct a randomized controlled trial substituting traditional forms of household energy (biomass for cooking and kerosene for lighting) with liquified petroleum gas (LPG) stoves/fuel and solar power (in areas marker for solar grids by the Government of Rwanda) in rural Rwanda. Eligible households (n=650) using traditional forms of energy will be recruited from eastern Rwanda. In each household, investigators will recruit either one adult female and one adult male or just one adult, and one child (aged 8-15 years). Following baseline health and exposure assessment, a randomized treatment arm (n=250 homes) will receive a full subsidy for LPG fuel and solar power, a control arm (n=250 homes) will continue to use traditional energy, and a random-subsidy arm (n=150 homes) will be randomized to a discounted price (at baseline and every 6-months) for solar and LPG in a pay-as-you-go (PAYG) service model (i.e., pre-pay a desired amount through mobile money). The random subsidy arm will then decide whether or not to cook with the discounted LPG or their traditional stove. Participants will be followed for 3 years with repeated measures of household air pollution (HAP) exposure (48-hour fine particulate matter (PM2.5) and black carbon (BC)), energy use, health, and preferences. Primary health endpoints include blood pressure (BP) in adults and lung-function growth in children; secondary endpoints include BP in children and lung-function change in adults. To complement the trial, the random-subsidy arm will generate policy-relevant information on causal relationships between energy costs, solar and LPG usage, and HAP exposures. The investigators propose 3 aims:

Aim 1. In an ITT framework, investigators will evaluate the effect of a household energy intervention on exposure to HAP and indicators of morbidity separately among Rwandan women, men, and children within n=500 households.

Aim 2. Using exposure-response modeling, investigators will characterize associations between exposure to HAP and indicators of morbidity separately among Rwandan women, men, and children within n=650 households (500 trial households + 150 random subsidy households).

Aim 3. Using a random-encouragement design, investigators will investigate causal relationships between randomized energy costs, measured energy usage, and estimated exposure to HAP among n=400 households (150 random subsidy households + 250 full subsidy treatment arm households).

ELIGIBILITY:
Inclusion Criteria:

This research will recruit and enroll 650 households (250 households in the full subsidy arm; 250 households in the control arm; 150 households in the discount subsidy arm).

The household level inclusion criteria is as follows:

* Home resides in the study area of Isangano and Karambi
* Uses biomass as primary cooking fuel
* Either both an adult male (at least 18 years old) and female (at least 18 years old), or just one adult (at least 18 years old), head(s) of household willing to consent and at least one child between 8 and 15 years of age willing to assent; We will recruit the younger child in families with more than one child between 8-15 years of age. We will also confirm the child is living at home throughout the year and not attending boarding school elsewhere.
* No commercial cooking
* No smoking in the household

Additional participant level inclusion is as follows:

* Not planning to move in 3-year timeframe
* Not currently pregnant (females); Note: If the female becomes pregnant during the study she will not be able to participate in any visits that occur during her pregnancy but she will be able to participate after she has given birth. However, if there is another adult in the household then this will not preclude the other two people (i.e., the other adult and the child) from continuing to participate throughout that time.

Exclusion Criteria:

The household level exclusion criteria is as follows:

* Home resides outside the study area
* Uses clean fuel as primary cooking fuel
* Participants outside the age ranges: Adult male (at least 18 years old) and female (at least 18 years old) heads of household willing to consent and at least one child between 8 and 15 years of age willing to assent
* Conducts commercial cooking
* Smoking members of the household

Additional participant level exclusion is as follows:

* Planning to move in 3-year timeframe
* Currently pregnant (females)

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1680 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2025-08-22 (Actual)

PRIMARY OUTCOMES:
Change in systolic blood pressure (adults) | Blood pressure will be measured approx. every 6 months for the 3-year follow-up period
Spirometry (children): FEV1 trajectory | Spirometry will be measured approx. every 6 months for the 3-year follow-up period
Spirometry (children): FVC trajectory | Spirometry will be measured approx. every 6 months for the 3-year follow-up period

SECONDARY OUTCOMES:
Change in systolic blood pressure (children) | Blood pressure will be measured approx. every 6 months for the 3-year follow-up period
Change in diastolic blood pressure (children) | Blood pressure will be measured approx. every 6 months for the 3-year follow-up period
Spirometry (children): FEV1/FVC trajectory | Spirometry will be measured approx. every 6 months for the 3-year follow-up period
Spirometry (children): FEF25-75 trajectory | Spirometry will be measured approx. every 6 months for the 3-year follow-up period
Spirometry (children): PEF trajectory | Spirometry will be measured approx. every 6 months for the 3-year follow-up period
Change in diastolic blood pressure (adults) | Blood pressure will be measured approx. every 6 months for the 3-year follow-up period
Spirometry (adults): FEV1 change | Lung function will be measured approx. every 1 year for the 3-year follow-up period (adults).
Spirometry (adults): FVC change | Lung function will be measured approx. every 1 year for the 3-year follow-up period (adults).
Spirometry (adults): FEV1/FVC change | Lung function will be measured approx. every 1 year for the 3-year follow-up period (adults).
Spirometry (adults): FEF25-75 change | Lung function will be measured approx. every 1 year for the 3-year follow-up period (adults).
Spirometry (adults): PEF change | Lung function will be measured approx. every 1 year for the 3-year follow-up period (adults).

CONTACTS AND LOCATIONS:
Locations (1):
- Field site in Rwanda (Isangano and Karambi), Ndego, Eastern Province, Rwanda

IPD SHARING:
Plan to Share IPD: Undecided